CLINICAL TRIAL: NCT01109615
Title: Phase II Study of Pemetrexed and Gemcitabine for Treatment Resistant Patients With Metastatic Colorectal Cancer and KRAS Mutations
Brief Title: Pemetrexed and Gemcitabine for Treatment Resistant Patients With Metastatic Colorectal Cancer and KRAS Mutations
Acronym: PG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lacking effect of treatment
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2010-018700-90
Record Dates: First submitted 2010-04-20; First posted 2010-04-23 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Metastatic colorectal cancer; Treatment resistant; Chemotherapy refractory; KRAS mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed — 400 mg/m2 on day 1 of a 3 weeks cycle
Drug: Gemcitabine — 1000 mg/m2 intravenously on day 1 and 8 of a 3 weeks cycle

SUMMARY:
This study aims to investigate the efficacy and safety of the combination of pemetrexed and gemcitabine in heavily pre-treated, chemotherapy resistant colorectal cancer patients with KRAS mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma in colon or rectum
* Age >18
* Metastatic colorectal cancer progressed after chemotherapy regimens containing fluoropyrimidines, oxaliplatin and irinotecan.
* KRAS mutation in primary tumour or metastasis.
* Measurable disease according to RECIST
* ECOG performance status 0, 1 or 2
* Adequate function of liver, kidneys and bone marrow measured by biochemistry (max. 2 weeks before enrolment)
* EDTA clearance: Uncorrected GFR > 45 ml/min.
* Neutrophilocytes ≥1.5 x 10^9/l, leukocytes ≥3.0 x 10^9/l, thrombocytes ≥100x10^9/l
* ALAT ≤ 3 x upper normal value (ULN), bilirubin ≤ 3 x upper normal value, Aptt and INR normal (or 2-3 at AC treatment). (ALAT and basic phosphatase ≤ 5 x upper normal value in case of liver metastases).
* Blood samples and paraffin embedded tissue from primary tumour and/or metastases for translational research.
* Fertile men and women (women <2 year after last menstruation) must use efficient birth control.
* Signed informed consent.

Exclusion Criteria:

* Clinically significant other concurrent disease making the patient unfit for participation in the study according to the investigator.
* Other malignant disease within 5 years prior to study enrolment, except from planocellular and basal cell carcinomas in the skin or carcinoma-in-situ cervix.
* Other experimental treatment within 30 days prior to treatment start.
* Pregnant or breastfeeding women.
* Clinical or radiological signs of CNS metastases.
* Planned radiation of target lesions.
* Concurrent vaccination against yellow fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Response rate | Assessed every 3 weeks by CT and/or MR scan and evaluated according to RECIST 1.1. Up to 12 months.

SECONDARY OUTCOMES:
Progression free survival | Every 3 months until progression or death. Up to 12 months.
Overall survival | 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark